CLINICAL TRIAL: NCT02234362
Title: Vortioxetine for Menopausal Depression and Associated Symptoms
Brief Title: Vortioxetine for Menopausal Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Marlene P. Freeman, MD, Associate Director, Center for Women's Mental Health, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P001812
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Depression; Menopause; Vasomotor Disturbance; Hot Flashes; Sleep
MeSH Terms: conditions — Depression; Hot Flashes | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open-label vortioxetine (Experimental): flexible-dose vortioxetine of 5-20 mg depending on tolerability
  Interventions: Drug: vortioxetine

INTERVENTIONS:
Drug: vortioxetine — Eligible subjects will initiate the treatment with 5 mg/day for two days and then 10 mg/day starting on Day 3. The dosage may be increased from 10 mg/day to 15 mg/day at Visit 2 or Visit 3. At Visit 4, the dosage may again be increased from 10 to 15 mg/day or from 15 to 20 mg/day, based on patient response and tolerability.
  Other Names: Trintellix

SUMMARY:
The broad goal of this study was to examine the efficacy and tolerability of vortioxetine (flexible dose) for the treatment of major depressive disorder (MDD) in symptomatic women around the menopausal transition. We hypothesized that an eight-week treatment with vortioxetine would promote a significant improvement of depression symptoms and other menopause-related physical symptoms.

DETAILED DESCRIPTION:
Forty-seven peri- and postmenopausal women were enrolled in this open-label study. This was an 8-week intervention using open-label vortioxetine with flexible dose between 5-20 mg, dependent on participant response and tolerability. In addition to assessment of depressive symptoms, improvement of menopause-related physical and emotional symptoms that occur with MDD, including vasomotor symptoms, cognition, fatigue, anxiety, sleep complaints, and quality of life, were also examined.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 40-62 years who are perimenopausal or early postmenopausal (within 5 years of the last menstrual period if not surgically postmenopausal), including:

   1. Perimenopausal women who have experienced changes in menstrual cycle frequency or duration, and/or physical symptoms indicative of menopausal transition, as determined by clinician
   2. Women who are using the Mirena Intrauterine Device (IUD), with Follicle-stimulating hormone (FSH) level > 20 milli-International unit/ml (mIU/mL)
2. Women meeting Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) criteria for major depression (assessed by the Mini International Neuropsychiatric Interview - M.I.N.I.)
3. MADRS scores of at least 20 at baseline visit
4. Women with significant menopause-related physical symptoms, indicated by any of the following criteria:

   1. Greene Climacteric Scale total scores > 20;
   2. Greene Climacteric Scale sub-score for vasomotor symptoms >3;
   3. 14 or more bothersome hot flashes per week (self-reported).
5. Signed informed consent.

Exclusion Criteria:

1. Pregnancy (determined by urine pregnancy test), intending pregnancy, or breast feeding.
2. Women whose primary diagnosis is Panic Disorder, Obsessive Compulsive Disorder (OCD), Generalized Anxiety Disorder (GAD), Seasonal Affective Disorder (SAD), or any other Axis I pathology active within 6 months prior to screening visit (except for specific phobias). Anxiety disorders are allowable if secondary to MDD as the primary diagnosis.
3. History of or current mania/hypomania, psychosis, or bipolar disorder
4. Regular treatment with an Selective Serotonin Reuptake Inhibitor (SSRI) or Selective Norepinephrine Reuptake Inhibitors (SNRI) within 2 months prior to screening visit
5. Serious suicidal ideation or intent
6. Women who have used psychoactive or centrally acting medications within 2 weeks prior to study screening
7. Women who have received hormonal intervention within 1 month prior to study entry
8. Known hypersensitivity to vortioxetine or any of the inactive ingredients
9. Treatment with a monoamine oxidase inhibitor (MAOI) within 14 days of randomization or potential need to use an MAOI during the study or within 21 days of discontinuation of study drug
10. Treatment with linezolid or intravenous methylene blue
11. Patients with severe hepatic impairment
12. Uncontrolled hypertension (>160/90 mmHg)
13. Resting heart rate >110/minute
14. Any current severe or unstable medical illness
15. Not using a medically approved method of birth control, if sexually active and not 12 or more months since last menstrual period
16. Drug or alcohol abuse in the past 1 year
17. Use of any disallowed medications (specified in the Excluded Concomitant Medication section below)
18. Concurrent enrollment in another clinical trial

Excluded Concomitant Medications:

* Selective estrogen-receptor modulators (SERMs)
* Hormone replacement therapy
* Hormonal contraceptives, excluding Mirena IUD
* Natural menopause supplements
* Episodic sleep medications (chronic, regular, stable-dose benzodiazepines are allowed)
* Antidepressants
* Phytoestrogens
* Soy-based medications
* Steroids
* Anorectics, appetite depressants

Ages: 40 Years to 62 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2015-06-12 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2016-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene P Freeman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bang-Andersen B, Ruhland T, Jorgensen M, Smith G, Frederiksen K, Jensen KG, Zhong H, Nielsen SM, Hogg S, Mork A, Stensbol TB. Discovery of 1-[2-(2,4-dimethylphenylsulfanyl)phenyl]piperazine (Lu AA21004): a novel multimodal compound for the treatment of major depressive disorder. J Med Chem. 2011 May 12;54(9):3206-21. doi: 10.1021/jm101459g. Epub 2011 Apr 12. PMID 21486038
- [Background] Bromberger JT, Assmann SF, Avis NE, Schocken M, Kravitz HM, Cordal A. Persistent mood symptoms in a multiethnic community cohort of pre- and perimenopausal women. Am J Epidemiol. 2003 Aug 15;158(4):347-56. doi: 10.1093/aje/kwg155. PMID 12915500
- [Background] Loprinzi CL, Kugler JW, Sloan JA, Mailliard JA, LaVasseur BI, Barton DL, Novotny PJ, Dakhil SR, Rodger K, Rummans TA, Christensen BJ. Venlafaxine in management of hot flashes in survivors of breast cancer: a randomised controlled trial. Lancet. 2000 Dec 16;356(9247):2059-63. doi: 10.1016/S0140-6736(00)03403-6. PMID 11145492
- [Background] Pehrson AL, Cremers T, Betry C, van der Hart MG, Jorgensen L, Madsen M, Haddjeri N, Ebert B, Sanchez C. Lu AA21004, a novel multimodal antidepressant, produces regionally selective increases of multiple neurotransmitters--a rat microdialysis and electrophysiology study. Eur Neuropsychopharmacol. 2013 Feb;23(2):133-45. doi: 10.1016/j.euroneuro.2012.04.006. Epub 2012 May 20. PMID 22612991
- [Background] Pehrson AL, Sanchez C. Serotonergic modulation of glutamate neurotransmission as a strategy for treating depression and cognitive dysfunction. CNS Spectr. 2014 Apr;19(2):121-33. doi: 10.1017/S1092852913000540. Epub 2013 Aug 1. PMID 23903233

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements in the greater Boston metropolitan area.
Period: Overall Study
Arm/Group | Open-label Vortioxetine
Started | 47
Received at Least One Dose of Medication | 27
Completed | 21
Not Completed | 26
Not completed — Not eligible after first screening visit | 17
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 27
Highest Level of Education [Count of Participants; unit: Participants]
  Some high school | 2
  High school or received GED | 7
  Vocational/training school after high school | 2
  Some college or Associate Degree | 8
  Graduated college (BA, BS) | 7
  Master's Degree | 1
  Doctoral Degree (PhD, MD, etc.) | 0
Employment [Count of Participants; unit: Participants]
  Full-or part-time work | 7
  Homemaker | 2
  Disabled | 3
  Not working, unemployed | 10
  Student | 0
  Volunteer | 1
  Retired | 2
  Temporary work | 2
Marital Status [Count of Participants; unit: Participants]
  Married | 6
  Separated/divorced/widowed | 8
  Never married/single | 13
  Decline to answer | 0
Menopausal Status [Count of Participants; unit: Participants]
  Perimenopausal | 13
  Naturally postmenopausal | 12
  Surgically postmenopausal | 2
Past hormone therapy use [Count of Participants; unit: Participants]
  Used hormone therapy in the past | 4
  Never used hormone therapy in the past | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale Score (MADRS) at Week 8 (Visit 5)
Description: The efficacy of vortioxetine for trea-ting depressive symptoms was measured by mean change in Montgomery-Asberg Depression Rating Scale (MADRS) depression score from Baseline (Visit 1) to Week 8 (Visit 5). The MADRS score was assessed at every study visit (Visits 1-5). Participants were considered to have responded to vortioxetine if their MADRS score was reduced by 50% or more from baseline to the end of treatment, and to be in remission if their final MADRS score was less than 10. Higher MADRS score indicates more severe depression. The overall MADRS score ranges from 0 to 60.
Time Frame: Baseline and Week 8 (Visit 5)
Population: The analyzable population includes all 24 participants who initiated medication treatment and returned for at least one assessment after starting vortioxetine. A last observation carried forward (LOCF) analysis was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 24
units on a scale | -22.8 (8.4)

2. Secondary Outcome: Change From Baseline in Vasomotor Symptoms (VMS) Frequency During Daytime at Week 8 (Visit 5)
Description: Vasomotor symptoms (VMS) were tracked and quantified prospectively using a daily hot flash diary. The hot flash diary was adapted from a 7-day self-report tool for vasomotor symptoms originally developed by the North Central Cancer Treatment Group (NCCTG). The diary asks for the subject to log number of hot flashes during the day and night, severity of hot flashes during day and night, and how bothersome the hot flashes were during day and night.
Time Frame: Baseline and Week 8 (Visit 5)
Population: The analyzable population includes all participants who initiated treatment with vortioxetine and returned for at least one assessment after study medication initiation who also reported having hot flashes at baseline.
Measure: Mean (Standard Deviation); unit: hot flashes per day
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 23
hot flashes per day | -1.33 (1.51)

3. Secondary Outcome: Change From Baseline in Vasomotor Symptoms (VMS) Severity During Daytime at Week 8 (Visit 5)
Description: Vasomotor symptoms (VMS) were tracked and quantified prospectively using a daily hot flash diary. The hot flash diary was adapted from a 7-day self-report tool for vasomotor symptoms originally developed by the North Central Cancer Treatment Group (NCCTG). The diary asks for the subject to log number of hot flashes during the day and night, severity of hot flashes during day and night, and how bothersome the hot flashes were during day and night.
  Severity of VMS:
  The range of scores for severity of VMS is 0-2, with higher scores indicating greater severity. 0=mild, 1=moderate, 2=severe
Time Frame: Baseline and Week 8 (Visit 5)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 23
units on a scale | -0.28 (0.43)

4. Secondary Outcome: Change From Baseline in Vasomotor Symptoms (VMS) Frequency During Nighttime at Week 8 (Visit 5)
Description: as for outcome 2
Time Frame: Baseline and Week 8 (Visit 5)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hot flashes per night
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 23
hot flashes per night | -1.15 (1.25)

5. Secondary Outcome: Change From Baseline in Vasomotor Symptoms (VMS) Severity During Nighttime at Week 8 (Visit 5)
Description: as for outcome 3
Time Frame: Baseline and Week 8 (Visit 5)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 23
units on a scale | -0.27 (0.37)

6. Secondary Outcome: Change From Baseline in Cognitive and Physical Functioning Questionnaire (CPFQ) Score at Week 8 (Visit 5)
Description: Cognition and physical functioning was measured by self-report responses to Cognitive and Physical Functioning Questionnaire (CPFQ).The range of scores is from 7-42. Higher scores indicate lower cognitive and executive functioning.
Time Frame: Baseline and Week 8 (Visit 5)
Population: The analyzable population includes all participants who initiated treatment with vortioxetine and returned for at least one assessment after study medication initiation.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 24
units on a scale | -13 [-15 to -7]

7. Secondary Outcome: Change From Baseline in Beck Anxiety Inventory (BAI) Score at Week 8 (Visit 5)
Description: Anxiety was measured by self-report responses to Beck Anxiety Inventory (BAI). It is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults. Several studies have found the Beck Anxiety Inventory to be an accurate measure of anxiety symptoms in children and adults. Higher scores on the BAI indicate more anxiety symptoms. The range of BAI scores is from 0 to 63, with 0-9=Minimal anxiety, 10-16=Mild anxiety, 17-29=Moderate anxiety, and 30-63=Severe anxiety.
Time Frame: Baseline and Week 8 (Visit 5)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 24
units on a scale | -7 [-12.5 to -0.5]

8. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) Score at Week 8 (Visit 5)
Description: Sleep quality and disturbances during the past month were assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI also incorporates daytime functioning into the total score. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. The range of scores is 0-21.
Time Frame: Baseline and Week 8 (Visit 5)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 24
units on a scale | -5 [-7.5 to -2.5]

9. Secondary Outcome: Change From Baseline in Menopause Specific Quality of Life (MENQOL) Score at Week 8 (Visit 5)
Description: Quality of life, menopause-specific, is assessed by the Menopause Specific Quality of Life (MENQOL).
  The MENQOL is self-administered and consists of a total of 29 items in a Likert-scale format. Each item assesses the impact of one of four domains of menopausal symptoms, as experienced over the last month: vasomotor (items 1-3), psychosocial (items 4-10), physical (items 11-26), and sexual (items 27-29). Items pertaining to a specific symptom are rated as present or not present, and if present, how bothersome on a zero (not bothersome) to six (extremely bothersome) scale. Means are computed for each subscale by dividing the sum of the domain's items by the number of items within that domain. Non-endorsement of an item is scored a "1" and endorsement a "2", plus the number of the particular rating, so that the possible score on any item ranges from 1-8. Total score also ranges from 1-8. Higher scores indicate that menopause symptoms are more bothersome.
Time Frame: Baseline and Week 8 (Visit 5)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 24
units on a scale | -1.74 [-2.61 to -1.30]

10. Secondary Outcome: Change From Baseline in Clinical Global Impression-Fatigue (CGI-F) Scale Score at Week 8 (Visit 5)
Description: Fatigue symptoms were assessed by the Clinical Global Impression-Fatigue (CGI-F) scale.The CGI-F is a single item global assessment scales to specifically evaluate symptoms of fatigue. Higher scores indicate more fatigue symptoms. The range of scores is from 0-7.
Time Frame: Baseline and Week 8 (Visit 5)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 24
units on a scale | -1 [-2.5 to 0]

11. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Scale Score at Week 8 (Visit 5)
Description: Severity of illness was assessed by the Clinical Global Impression-Severity (CGI-S) Scale. The CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. The range of scores is 0-7. Higher scores indicate greater severity of illness.
Time Frame: Baseline and Week 8 (Visit 5)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 24
units on a scale | -1 [-2.5 to -1]

12. Secondary Outcome: Change From Baseline in Pain Assessment (PEG) Score at Week 8 (Visit 5)
Description: Pain symptoms were assessed by the Pain Assessment (PEG). The PEG is a three-item scale assessing pain intensity and interference. A higher score indicates more pain symptoms. The range of scores is from 0 to 30.
Time Frame: Baseline and Week 8 (Visit 5)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 24
units on a scale | -4 [-9.5 to 0]

13. Secondary Outcome: Change From Baseline in Greene Climacteric Scale (GCS) Score at Week 8 (Visit 5)
Description: Menopause related symptoms were assessed using the Greene Climacteric Scale (GCS). The Greene Scale provides a brief measure of menopause symptoms. It can be used to assess changes in different symptoms, before and after menopause treatment. Three main areas are measured:
  1. Psychological (items 1-11). 2. Physical (items 12-18). 3. Vasomotor (items 19, 20).
  A higher score indicates that menopause symptoms are more bothersome. The range of scores is from 0 to 63.
Time Frame: Baseline and Week 8 (Visit 5)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 24
units on a scale | -18.5 [-25 to -13.5]

14. Secondary Outcome: Change From Baseline in Digit Symbol Substitution Test (DSST) Score at Week 8 (Visit 5)
Description: Processing speed, working memory, visuospatial processing and attention was assessed by the Digit Symbol Substitution Test (DSST).
  The DSST test requires the examinee to transcribe a unique geometric symbol with its corresponding Arabic number. The examinee is initially shown a key containing the numbers from 1 to 9. Under each number there is a corresponding geometric symbol. The examinee is then shown a series of boxes containing numbers in the top boxes, and blank boxes below them. After a short practice trial, they are then asked to copy the corresponding geometric symbol under each number. The raw score is the number of correct items completed within the prescribed time limit. Higher scores indicate faster processing speed, working memory, and visuospatial processing and attention. The range of scores is 0-63.
Time Frame: Baseline and Week 8 (Visit 5)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Open-label Vortioxetine
Number analyzed (Participants) | 24
units on a scale | 8.5 [4.5 to 15.5]

ADVERSE EVENTS:
Time Frame: Adverse event data were assessed from baseline through Week 8 (Visit 5) of the study. At each study visit, physician investigators prompted the participant to report any occurrences of health problems other than usual menopause related symptoms. Any serious or non-serious adverse events were recorded in the participant's study binder at each examination.
Arm/Group | Open-label Vortioxetine
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 21/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Vortioxetine (N=27)
Nausea (General disorders) | 13
Headaches (Nervous system disorders) | 7
Dry mouth (General disorders) | 5
Vomiting (Gastrointestinal disorders) | 3
Increased thirst (General disorders) | 2
Dizziness (General disorders) | 2
Stomach cramps (Gastrointestinal disorders) | 1
Mild rash (Skin and subcutaneous tissue disorders) | 1
Abdomen tenderness (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
Numbness (Nervous system disorders) | 1
Restlessness (General disorders) | 1
Disrupted sleep (General disorders) | 1
Difficulty falling asleep (General disorders) | 1
Decreased appetite (General disorders) | 1
Increased appetite (General disorders) | 1
Hair loss (Skin and subcutaneous tissue disorders) | 1
Increased fatigue (General disorders) | 1
Decreased libido (Reproductive system and breast disorders) | 1
Anorgasmia (Reproductive system and breast disorders) | 1
Palpitations (Cardiac disorders) | 1
Edginess (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Blurred vision (Eye disorders) | 1
Increased Anxiety (Psychiatric disorders) | 1

LIMITATIONS AND CAVEATS:
* lack of control group (important given that previous VMS medication trials have indicated modest placebo response rates, and it is difficult to determine whether the side effects are associated with the medication)
* small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No